CLINICAL TRIAL: NCT06330870
Title: Evaluation of Brain Metastasis Development Mechanism in Patients With Breast Cancer With Brain Metastasis(BCBM)
Brief Title: Brain Metastasis Development Mechanism in BCBM Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JI-YEON, KIM, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BCBM_Breast
Record Dates: First submitted 2024-02-06; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Brain Metastasis
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGS/TME evaluation (Experimental): This is not intervention clinical trial design. We explore whole genome sequencing and tumor microenvironment evaluation for brain metastasis specimen in breast cancer patients.
  Interventions: Procedure: WGS/TME evaluation

INTERVENTIONS:
Procedure: WGS/TME evaluation — WGS/TME evaluation with blood and brain metastasis tissue during brain metastasis curative surgery

SUMMARY:
This study is the experimental study for brain metastasis development mechanism in patients with breast cancer with brain metastasis

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Brain metastasis curative surgery patient

Exclusion Criteria:

* Gamma Knife surgery patient

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial disease free survival | Months
  Time to new brain metastasis or brain metastasis progression from the brain surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ji-Yeon Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No